CLINICAL TRIAL: NCT06817941
Title: Enhancing Rehabilitation Outcomes in Cerebral Palsy Through Gamified Multidisciplinary Interventions: Integrating Speech and Upper Extremity Motor Therapy
Brief Title: Speech and Arm Combined Exergame
Acronym: SPACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Young Hwa Michelle Chang, Ph.D., CCC-SLP, Assistant professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2024001772
Record Dates: First submitted 2025-01-24; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy (CP); Dysarthria
Keywords: cerebral palsy; children; dysarthria; motor speech disorder; upper extremity; arm weakness; intervention; video games; fNIRS; neuroimaging; therapy; rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Dysarthria; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Speech only (Group 1) (Experimental): Participants in Group 1 will play three video games using their voice only.
  Interventions: Behavioral: Speech only
- Arm only (Group 2) (Experimental): Participants in Group 2 will play three video games using their impaired hand and arm only.
  Interventions: Behavioral: Hand/Arm only
- Speech/Arm combined (Group 3) (Experimental): Participants in Group 3 will play three video games using both voice and hand/arm.
  Interventions: Behavioral: Speech and arm combined

INTERVENTIONS:
Behavioral: Speech only — Participants will be using a computer-based speech therapy games at home to train their speech clarity for 8 weeks. While playing these games, a webcam will be recording the participant's speech loudness and mouth opening.
  Arms: Speech only (Group 1)
Behavioral: Hand/Arm only — Participants will be using a computer-based therapy games at home to train their hand and arm movement for 8 weeks. While playing these games, a motion detector will be used to measure how quickly and accurately the participants can move their fingers, wrist, and arm.
  Arms: Arm only (Group 2)
Behavioral: Speech and arm combined — Participants will be using a computer-based therapy games at home to train their speech clarity and hand/arm movement together for 8 weeks. While playing these games, a webcam will be recording the participant's speech loudness and mouth opening. A motion detector will also be used to measure how quickly and accurately the participants can move their fingers, wrist, and arm.
  Arms: Speech/Arm combined (Group 3)

SUMMARY:
The purpose of this study is to develop innovative home therapy games to train the weak arm and improve speech intelligibility (clarity) of children with hemiplegia from cerebral palsy. The investigators are exploring the effects of these therapy games and how they change the children's speech, hand movement, and brain activation.

15 children who are 8-17 years old will be recruited for this study. These children should have a diagnosis of cerebral palsy, mild to moderate speech issues but use speech as the primary mode of communication, mild to moderate movement difficulty and muscle spasticity, adequate hearing (pass a hearing screening), and be able to follow simple task-related directions.

Children who have severe vision impairment that limits the child's ability to interact with the entire computer screen, have severe arm weakness so they cannot move their arm enough to interact with the computer games, have severe increase in tone in their weak arm, or have difficulty following instructions or paying attention to computer video games for at least 10 minutes cannot participate in this study.

The therapy games will take 8 weeks to finish at home. Each child will play these games for 30 minutes each day, 5 days per week.

In addition, children will come to the lab 4 times for speech and hand movement assessment: (1) 1st assessment takes place immediately before the child start to play the video games. (2) 2nd assessment takes place 4 weeks (midpoint) after the child starts to play the games. (3) 3rd assessment takes place immediately after the video games are finished. (4) 4th assessment takes place 6 weeks after the video games are finished.

Each assessment should take about 2 hours to complete in the Rutgers movement lab or at Rutgers SLP Clinic.

A total of 15 children will take part in this research study. The research will last for 2 years overall.

DETAILED DESCRIPTION:
In recent decades, rigorous treatment utilizing the principles of motor learning and activity-dependent neuroplasticity have shown significant improvement in speech and upper extremity (UE) function in children with cerebral palsy (CP). While intensive motor treatment can provide significant therapeutic benefits, it is often difficult for children to participate and complete such therapy, especially when they find the process to be tedious or lack immediate feedback and tracking of improvement over time. The need to maximize engagement during therapy is thus pivotal to ensure that treatment is both effective and sustainable. To this end, gamified therapy may be ideal, as it has been well-documented in literature to enhance not only targeted motor functions during UE therapy but also participation and motivation in children. Furthermore, combining speech and UE in a multidisciplinary gamified therapy may provide benefits to many children with CP who have concomitant impairment of speech and UE. Due to the neurological similarities underlying speech production and hand/arm movement execution, synergistic effects may be expected when treating both domains simultaneously. Research on this clinically significant topic deserves attention and further examination.

Specifically, in this proposed study, the following aims will be targeted:

Aim 1: Develop computer-based therapy games designed to improve speech intelligibility and UE function.

Aim 2: Evaluate the feasibility and effectiveness of a gamified multidisciplinary treatment method (i.e., combined speech and UE) and compare it to the independent effects of gamified speech and UE therapy.

Aim 3: Examine the potential overlap in the neural correlates of speech and UE movement as well as the post-treatment changes in these correlates under the combined versus independent conditions.

The goal of this project is to develop and evaluate the feasibility and effectiveness of a gamified multidisciplinary treatment for speech and UE, and to examine the underlying neural correlates of the two domains in response to treatment. This approach will enhance participation of children with CP and, consequently, the effectiveness of therapy aimed at improving speech intelligibility and UE function. Furthermore, the games that will be developed can be part of a home-based therapy system and thus used in telerehabilitation to provide treatment to a much greater number of children. The impact of these research goals is crucial to refine therapeutic approaches and tailor them to meet the specific needs of children with CP, ultimately aiming to increase the children's independence and improve their quality of life.

Cerebral Palsy (CP) is the leading cause of motor impairment in children. Approximately 1 in 345 children in the United States have CP. It is a heterogeneous, nonprogressive, and lifelong disorder, with many children presenting with the motor speech disorder of dysarthria as well as sensorimotor issues of the upper limb. The intelligibility reductions in dysarthria, along with the sensorimotor issues affecting the upper extremities, often limit these children's ability to communicate and perform activities of daily living (ADLs). This may negatively impact social development, reduce their quality of life, and result in social isolation or depression. Therefore, therapeutic exercises targeting improvement in speech and UE are essential for children with CP throughout life as they reach new developmental milestones and functional demands.

Gamified upper extremity (UE) and speech treatment for children with CP:

Positive effects of gamified therapy have been documented in children with CP for UE training. Training using computer-based games showed greater recovery of upper extremity function compared to traditional therapies in young people with CP in multiple studies, but that most studies were of lower quality and design. In addition to UE limitations, more than 50% of children with CP present with a motor speech disorder of dysarthria, which can negatively impact speech intelligibility and create a barrier to communication. Therefore, improving intelligibility is also a fundamental goal of speech intervention for this population.

This research seeks to develop computer-based therapy games to train the UE and speech in children with CP. The UE training component will focus on fine motor activities needed to perform activities of daily living. The speech training component leverages the intelligibility benefits of an intensive speech treatment method for children with CP (i.e., Speech Intelligibility Treatment; SIT).

Multidisciplinary treatment:

Speech and UE therapy will be integrated into a multidisciplinary gamified treatment to investigate the benefits of combined speech and UE training. Such combined treatment may be effective because speech and arm motions are linked together behaviorally, neurologically, and developmentally. Furthermore, since children with CP often receive multiple types of therapies together, a multidisciplinary goal-directed treatment that targets specific movement skills in speech and UE will be clinically and practically applicable. Such co-treatment will facilitate more seamless care, rather than speech-language and mobility gains being made in a fragmented manner. Finally, both speech and arm motor training follow similar motor learning principles, which state that incorporating contextual interference during skilled motor training may lead to greater retention of learned skills. For example, improvement in fine motor skills may transfer to enhancements in motor control elsewhere, including the orolingual muscles of articulation. Combining speech and UE motor training may, therefore, allow for interdisciplinary skill transfer, which will result in more enduring benefits and the retention of acquired abilities.

Neural correlates of speech and UE movement changes:

Execution of UE movement recruits activation of cortical areas in the primary sensorimotor system, premotor areas, and executive networks such as the parietal cortex and prefrontal cortex. Similarly, speech execution recruits areas in the sensorimotor and frontoparietal cortices. This overlap in cortical resources raises important questions about whether training UE movement and speech simultaneously would increase activations of these overlapping cortical areas or decrease them due to competition. Furthermore, questions of whether simultaneous training leads to a change in the activation pattern of all the cortical resources remain unanswered. We aim to answer these questions by utilizing the fNIRS technology to compare the neural changes as a function of treatment.

This study will advance the field's knowledge of combined speech and UE therapy, and how such multidisciplinary treatment can be beneficial to children with CP. Successful completion of this research may ultimately increase the children's independence and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosis of CP
* (2) age between 8-17 years (i.e., pediatric age)
* (3) use speech as the primary mode of communication
* (4) mild to moderate dysarthria
* (5) Manual Ability Classification System (MACS) level I to III
* (6) Gross Motor Function Classification System (GMFCS) level I to IV
* (7) mild to moderate muscle spasticity of the arm with a Modified Tardieu Scale of 0-3
* (8) pass bilateral pure-tone hearing screening at 25 dB HL (at 500, 1000, 2000, and 4000 Hz)
* (9) able to follow simple task-related directions, including repeating short phrases.

Exclusion Criteria:

* (1) severe vision impairment that limits the child's ability to interact with the entire computer screen
* (2) dyskinetic CP or spastic diplegia
* (3) English is not their first or primary language.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Intelligibility measures | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  To assess the word and sentence intelligibility changes in the participating children with CP. Once the child participants' data are collected, adult listeners will come to the Rutgers SLP Clinic to assess speech changes in these children. Each listener will spend approximately 30 minutes to one hour listening to the children's speech (words and sentences) and type on a laptop what they heard. They will also indicate how easy or difficult the utterance was to understand using a visual analog scale on the laptop. The anchor points provided on the scale will be: difficult to understand (score = 0) to easy to understand (score = 100). Each listener will provide their rating by sliding a pointer on this scale between the two anchor points. The words and sentences that the listeners listen to are audio recordings collected during the child participants' four assessment sessions (pre-treatment, mid-treatment, post-treatment, and retention).
Melbourne Assessment 2 | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  MA2 is a 14 item criterion-referenced test for evaluating four elements of upper limb movement quality in children with a neurological impairment

SECONDARY OUTCOMES:
Speech rate | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  The speed at which the participant can articulate a word (syllables per second) or a sentence (words per second)
Vowel space area | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  Area of oral aperture during speech, measured with four American English corner vowels
Sound pressure level | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  Loudness of speech, measured in dB
FOCUS questionnaire | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  Social communication questionnaire that examines how the participants' use of speech changed after treatment
Box and Block test (BBT) | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  BBT is a standardized activity level test used to measure the gross manual dexterity. The subject is given 60 seconds to move as many blocks as possible over a partition to the other, using one hand.
Fingers range of motion | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  The Hand Open Range value is calculated by measuring the difference in the average distance between the fingertips and the center of the palm across all four fingers in these two positions.
Wrist range of motion | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  The participant extends and flexes their wrist against gravity with their forearm in a fixed position. Angular difference between these two positions is reported as the wrist pitch range.
Forearm range of motion | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  The participant moves and holds their hand in pronation and supination with their elbow fixed.
Speed of fingers open/close | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  Measure how many times the participants can open and close fingers in 5 seconds.
Speed of wrist flexion/extension | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  Measure how many times the participants can move the wrist up and down (flex, extend) in 5 seconds
Speed of forearm pronation/supination | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  Measure how many times the participants can rotate their forearm in 5 seconds
Accuracy of finger open/close | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  The participant attempts to trace an irregular wave which moves on the screen from left to right at a constant speed. Accuracy is calculated as the root mean square error between the cursor position and the corresponding target point on the wave.
Accuracy of wrist flexion/extension | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  The participant controls a cursor that moves up and down by flexing and extending their wrist. Task and accuracy values are calculated.
Accuracy of forearm pronation/supination | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  The participant controls a cursor that moves up and down by pronating and supinating their hand. Task and accuracy calculations were performed.
Handheld Dynamometry | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  Grip strength measured with hand dynamometry
CP-QOL | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  Quality of life measure for person with CP
fNIRS | Pre-treatment (1-2 weeks before treatment), mid-treatment (4 weeks after treatment begins), post-treatment (immediately after treatment ends at 8 weeks), 6-week retention (6 weeks after treatment ends)
  fNIRS will be used as a measure of hemodynamic activation during speech and hand/arm movement tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Young Hwa M Chang, PhD, CCC-SLP, Principal Investigator — Rutgers University
Locations (1):
- Rutgers School of Health Professions, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study, and therefore, we do not plan to share IPD.

REFERENCES:
- [Background] Levy ES, Chang YM, Hwang K, McAuliffe MJ. Perceptual and Acoustic Effects of Dual-Focus Speech Treatment in Children With Dysarthria. J Speech Lang Hear Res. 2021 Jun 18;64(6S):2301-2316. doi: 10.1044/2020_JSLHR-20-00301. Epub 2021 Mar 3. PMID 33656916